CLINICAL TRIAL: NCT03734133
Title: Electromyography Evaluation of the Impacts of Different Insoles in the Activity Patterns of the Lower Limb Muscles: A Cross-over Quasi-experimental Study
Brief Title: Electromyography Evaluation of the Impacts of Different Insoles in the Activity Patterns of the Lower Limb Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, César Calvo Lobo, Principal Investigator, Universidad de León
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMG_foot orthoses
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Electromyography; Muscles; Foot Orthoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Foot orthoses (Experimental): Different foot orthoses
  Interventions: Other: Foot insoles

INTERVENTIONS:
Other: Foot insoles — Different foot insoles of different hardness

SUMMARY:
The main objective of this research is to demonstrate that the use of insoles of different hardness in motorcycle riders may cause variations in the electromyographic activity of the lower limb muscles during the race. This study is a cross-over quasi-experimental study. Nine motorcycle riders were recruited. Electromyographic activity of the lower limb muscles is recorded under different insole types.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Motorcycle riders

Exclusion Criteria:

* Musculoskeletal conditions
* Neurological alterations
* Systemic diseases.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Superficial electromyography peak measured as percentage | Change from Baseline superficial electromyography peak at 5 minutes
  Superficial electromyography activity peak of the vastus lateralis muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No